CLINICAL TRIAL: NCT00655772
Title: A Randomized, Double Blind, Crossover, Placebo-Controlled Clinical Trial to Assess the Effects of a Mouthwash Containing Chlorine Dioxide on Oral Malodor
Brief Title: A Clinical Trial to Assess the Effects of a Mouthwash Containing Chlorine Dioxide on Oral Malodor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tokyo Medical and Dental University (Other)
Responsible Party: Kayoko Shinada/DDS, PhD, Dept. of Oral health promotion, Tokyo medical and dental university
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1_Shinada
Record Dates: First submitted 2008-03-28; First posted 2008-04-10 (Estimated); Last update posted 2008-04-10 (Estimated); Status verified 2008-03

CONDITIONS: Halitosis
Keywords: chlorine; dioxide; mouthwash; organoleptic; measurements; volatile; sulfur; compounds
MeSH Terms: conditions — Halitosis | interventions — chlorine dioxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Chlorine Dioxide — Experimental mouthwash (ClO2 Fresh®): 0.16% sodium chlorite (NaClO2) with an efficacy of 0.1% chlorine dioxide (ClO2),Placebo mouthwash: glycerin, mint oil and distilled water, contents are almost the same as those in the experimental mouthwash except ClO2.
  Other Names: ClO2 Fresh®

SUMMARY:
A mouthwash containing chlorine dioxide would be effective to reduce oral malodor.

DETAILED DESCRIPTION:
A randomized, double blind, crossover, placebo-controlled clinical trial was conducted among 15 healthy male volunteers, who were divided into 2 groups: experimental or control group. In the first test phase, the subjects in the experimental group were instructed to rinse with the mouthwash containing ClO2 and those in the control group with the placebo mouthwash without ClO2. In the second test phase after one week washout period, same procedure was conducted with the opposite mouthwashes. Oral malodor was evaluated at before rinsing, right after rinsing and follows up every 30 minutes till 4 hours with OM, and the concentrations of hydrogen sulfide (H2S), methyl mercaptan (CH3SH) and dimethyl sulfide ((CH3)2S) which are the main volatile sulfur compounds (VSCs) of human oral malodor were evaluated with GC.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of oral malodor
* Rinsing the mouthwash

Exclusion Criteria:

* oral malodor caused by foods

Ages: 19 Years to 38 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-02; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Oral malodor was evaluated at before rinsing, right after rinsing and follows up every 30 minutes till 4 hours with organoleptic measurements. | 4 hours

SECONDARY OUTCOMES:
Oral malodor was evaluated at before rinsing, right after rinsing and follows up every 30 minutes till 4 hours with the concentrations of 3 kinds gases of human oral malodor analyzing with gas chromatography. | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kayoko Shinada, DDS, PhD, Principal Investigator — Dept. of Oral health promotion, Tokyo medical and dental university
Locations (1):
- Dept. Oral health promotion, Tokyo medical and dental university, Yushima Bunkyo-ku, Tokyo, Japan

REFERENCES:
- [Derived] Shinada K, Ueno M, Konishi C, Takehara S, Yokoyama S, Kawaguchi Y. A randomized double blind crossover placebo-controlled clinical trial to assess the effects of a mouthwash containing chlorine dioxide on oral malodor. Trials. 2008 Dec 9;9:71. doi: 10.1186/1745-6215-9-71. PMID 19068114